CLINICAL TRIAL: NCT05513950
Title: A Phase Ib, Randomised, Double-blind, Placebo-controlled Study to Investigate the Safety, Tolerability, and Pharmacokinetics of an Intravenous Monoclonal Antibody (mAb) After Single Ascending Doses in Subjects Affected by Idiopathic Pulmonary Fibrosis.
Brief Title: A Study to Investigate the Safety, Tolerability, and Pharmacokinetics of Monoclonal Antibody (mAb) in Patients With IPF (SAD).
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLI-10067AA1-01
Record Dates: First submitted 2022-08-17; First posted 2022-08-24 (Actual); Results first posted 2025-08-14 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-07

CONDITIONS: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Intervention Model Description: Treatment with single dose escalation: 3 separate cohorts received 3 incremental doses of Investigational Medicinal Product (IMP). Each cohort started when the previous cohort was completed and the data were evaluated by the Safety Advisory Committee.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The Investigational Medicinal Product (IMP) was blinded for the participant, investigators, and the sponsor. At the study site an unblinded pharmacist (or designee) prepared the IMP and an unblinded clinical research associate checked the documents of the IMP preparation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Treatment (Experimental): A single intravenous (IV) dose of CHF10067
  Interventions: Biological: CHF10067 starting dose -- 1000mg (Cohort A); Biological: CHF10067 intermediate dose -- 2000mg (Cohort B); Biological: CHF10067 high dose -- 3000mg (Cohort C)
- Reference treatment (Placebo Comparator): A single dose of placebo (commercial source of 0.9% sodium chloride aqueous solution)
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: CHF10067 starting dose -- 1000mg (Cohort A) — Intravenous administration of a starting dose of the monoclonal antibody
  Arms: Test Treatment
Biological: CHF10067 intermediate dose -- 2000mg (Cohort B) — Intravenous administration of an intermediate dose of the monoclonal antibody
  Arms: Test Treatment
Biological: CHF10067 high dose -- 3000mg (Cohort C) — Intravenous administration of a high dose of the monoclonal antibody
  Arms: Test Treatment
Drug: Placebo — Intravenous administration of a physiological solution as placebo
  Arms: Reference treatment

SUMMARY:
Assess the safety of CHF10067 (study drug) and any side effects that might be associated with it. The study also evaluated how much of the study drug gets into the bloodstream and how long the body takes to remove it. The body's immune response to the study drug was evaluated.

Chiesi conducted this study in patients affected by idiopathic pulmonary fibrosis (IPF, a progressive and chronic lung disease). Chiesi performed this study to establish the drug doses that would be suitable for future studies (a dose finding study).

DETAILED DESCRIPTION:
The principal aim of this study was to obtain safety and tolerability data when CHF10067 was administered intravenously as single ascending doses to subjects with IPF (a progressive and chronic lung disease). This information, together with the pharmacokinetic (PK) and immunogenicity data is part of a dose finding efforts, for future clinical studies. The effect of CHF10067 on transglutaminase 2 (TG2) levels was also investigated as an exploratory endpoint.

A sequential group, single ascending dose design has been chosen for safety reasons because CHF10067 is in the early stages of clinical development and no data in the IPF population has been collected so far. In addition, sentinel dosing was used so that in each cohort 2 subjects (1 CHF10067 and 1 placebo) was administered at least 24 hours, before the remaining 6 subjects.

The study was double-blind and placebo-controlled to avoid bias in the collection and evaluation of data during its conduct. Placebo was chosen as the comparison treatment to assess whether any observed effects are treatment-related or reflect the study conditions.

ELIGIBILITY:
Inclusion Criteria:

* Subject's written informed consent obtained prior to any study-related procedure.
* Males or females, of any race, aged ≥ 40 years of age.
* Body weight ≥ 45 kg.
* Diagnosis of IPF as defined by current American Thoracic Society/European Respiratory Society/Japanese Respiratory Society/Latin American Thoracic Association guidelines. Diagnosis of IPF must be within the past 5 years prior to enrolment, and in the opinion of the Investigator, has been stable for at least 3 months.
* Subjects not receiving any IPF treatment (including subjects with previous use of antifibrotic treatment that has been stopped for at least 2 weeks prior to screening) or receiving well-tolerated standard of care approved treatments at a stable dose for at least 8 weeks prior to screening (nintedanib or pirfenidone) and it is anticipated the dose will remain unchanged throughout the study.
* Forced vital capacity (FVC) ≥ 50% of predicted and ratio of forced expiratory volume in the first second (FEV1)/FVC ≥ 0.7 at screening.
* Diffusing capacity of the lung for carbon monoxide (DLCO; corrected for haemoglobin) ≥ 35% at screening.
* Able to understand the study procedures and the risks involved.
* Male and Female subjects following contraceptive requirements detailed in the study protocol.

Exclusion Criteria:

* History of lower respiratory tract infection within 4 weeks prior to screening and up to Day 1 of the study.
* History of acute exacerbation of IPF within 3 months prior to screening and up to Day 1 of the study
* Active diagnosis of lung cancer or a history of lung cancer.
* Active cancer or a history of cancer (other than lung cancer) with less than 5 years disease free survival time (whether or not there is evidence of local recurrence or metastases).
* Infiltrative lung disease other than IPF
* Subjects exhibiting unhealed wounds or foot ulcers or have known history of wound healing complications.
* Chronic heart failure categorized as New York Heart Association Class II, III, or IV; clinical diagnosis of cor pulmonale requiring specific treatment; or severe pulmonary hypertension
* Currently receiving, or have received, a systemic corticosteroid, immunosuppressant, cytotoxic therapy, vasodilator therapy for pulmonary hypertension, or unapproved or investigational treatment for IPF within 4 weeks prior to screening or prior to randomization.
* Coronavirus disease-2019 (COVID-19) vaccine at least 7 days before dosing. Any systemic symptoms (e.g. myalgia, fever, chills, fatigue, etc.) after COVID-19 vaccine should subside at least 2 days before the Day 1 visit.
* Documented COVID-19 diagnosis within the last 4 weeks or which has not resolved within 7 days prior to screening or before treatment.
* Known intolerance and/or hypersensitivity to any of the excipients contained in the formulation or any other substance used in the study.
* History of allergic or anaphylactic reaction to human, humanised, chimeric, immunoglobulins (Igs), or murine monoclonal antibodies.
* Clinically relevant abnormal laboratory values (clinical chemistry and haematology) at screening suggesting an unknown disease and requiring further clinical investigation or which may impact the safety of the subject or the evaluation of the study results according to Investigator judgement. .
* Pregnant or lactating women.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2023-01-25 (Actual); Primary Completion 2024-06-17 (Actual); Study Completion 2024-06-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Spencer, Principal Investigator — Liverpool University Hospitals NHS Foundation Trust
Locations (9):
- PHI University Clinic of Pulmonology and Allergology, Skopje, North Macedonia
- Medical Center of Limited Liability Company "Arensia Exploratory Medicine", department of Clinical Trials, Kyiv, Ukraine
- United Kingdom (7):
  - Queen Elizabeth Hospital - NIHR Birmingham Clinical Research Facility - University Hospitals Birmingham NHS Foundation Trust, Birmingham
  - Royal Papworth Hospital NHSFT - Cambridge Biomedical Campus, Cambridge
  - University of Dundee, NHS Tayside - Ninewells Hospital & Medical School, Dundee
  - Interstitial Lung Disease Research - NHS Lothian - Royal Infirmary of Edinburgh,, Edinburgh
  - Liverpool Clinical Research Facility - Liverpool University Hospital Foundation Trust, Liverpool
  - Medicines Evaluation Unit - The Langley Building, Manchester
  - University Hospital Southampton - Department of Respiratory Medicine, Southampton

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: For the study, 52 male and female subjects were screened 3-28 days before randomization; of these, 27 subjects were screening failures. Overall, 25 subjects were randomized; of these 1 subject (CHF 10067 3000 mg) did not receive the study medication due to technical reasons.
Groups:
- CHF 10067 1000 mg (Test Treatment): A single intravenous (IV) dose of CHF10067
  CHF10067 starting dose: Intravenous administration of a starting dose of the monoclonal antibody
- CHF 10067 2000 mg (Test Treatment): A single intravenous (IV) dose of CHF10067
  CHF10067 intermediate dose: Intravenous administration of an intermediate dose of the monoclonal antibody
- CHF 10067 3000 mg (Test Treatment): A single intravenous (IV) dose of CHF10067
  CHF10067 high dose: Intravenous administration of a high dose of the monoclonal antibody
- Placebo: A single dose of placebo (commercial source of 0.9% sodium chloride aqueous solution)
  Placebo: Intravenous administration of a physiological solution as placebo
Period: Overall Study
Arm/Group | CHF 10067 1000 mg (Test Treatment) | CHF 10067 2000 mg (Test Treatment) | CHF 10067 3000 mg (Test Treatment) | Placebo
Started | 6 | 6 | 7 | 6
Completed | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 1 | 0
Not completed — Not treated due to technical reasons | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- CHF 10067 3000 mg (Test Treatment): A single intravenous (IV) dose of CHF10067
  CHF10067 high dose: Intravenous administration of an high dose of the monoclonal antibody
- Total: Total of all reporting groups
Arm/Group | CHF 10067 1000 mg (Test Treatment) | CHF 10067 2000 mg (Test Treatment) | CHF 10067 3000 mg (Test Treatment) | Placebo | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.7 (7.3) | 61.8 (8.0) | 58.7 (8.2) | 70.7 (4.1) | 63.0 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 5 | 0 | 8
  Male | 5 | 4 | 1 | 6 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 6 | 6 | 6 | 6 | 24
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 25.98 (2.17) | 30.23 (3.66) | 30.02 (4.18) | 27.80 (1.90) | 28.51 (3.42)
Smoking status at screening [Count of Participants; unit: Participants]
  Tobacco: Ex-smoker | 3 | 3 | 3 | 4 | 13
  Tobacco: Non-smoker | 3 | 3 | 3 | 2 | 11
  E-cigarettes: Ex-smoker | 0 | 0 | 0 | 0 | 0
  E-cigarettes: Non-smoker | 6 | 6 | 6 | 6 | 24
Duration of smoking [Mean (Standard Deviation); unit: years] — Population: Data available only for ex-smokers.
  years
    number analyzed (Participants) | 3 | 3 | 3 | 4 | 13
    (all) | 40.3 (7.8) | 33.7 (16.3) | 21.7 (5.7) | 24.5 (16.3) | 29.6 (13.5)
Number of pack-years [Mean (Standard Deviation); unit: pack-years] — Pack-year: is calculated by multiplying the number of packs of cigarettes smoked per day by the number of years the person has smoked. Population: Data available only for ex-smokers.
  pack-years
    number analyzed (Participants) | 3 | 3 | 3 | 4 | 13
    (all) | 18.60 (8.79) | 22.43 (18.60) | 20.00 (7.00) | 18.00 (13.98) | 19.62 (11.43)
Time since diagnosis [Median (Full Range); unit: years] | 1.25 [0.6 to 4.1] | 0.79 [0.3 to 4.1] | 1.21 [0.0 to 4.4] | 1.40 [0.2 to 4.6] | 1.00 [0.0 to 4.6]
Type of diagnosis [Count of Participants; unit: Participants] — Population: Results are provided for subjects with relevant diagnostic data.
  IPF=Idiopathic pulmonary fibrosis; HRCT=High-resolution computed tomography; UIP=Usual interstitial pneumonia;
  Participants
    UIP pattern on available HRCT scan prior to screening | 3 | 5 | 4 | 3 | 15
    Possible UIP pattern on available HRCT scan prior to screening: number analyzed (Participants) | 6 | 6 | 6 | 3 | 21
    Possible UIP pattern on available HRCT scan prior to screening | 0 | 0 | 0 | 0 | 0
    Probable UIP pattern on available HRCT scan prior to screening. IPF confirmation: YES | 3 | 1 | 2 | 3 | 9
    Probable UIP pattern HRCT scan prior to screening. Lung biopsy in accordance with HRCT: NA: number analyzed (Participants) | 3 | 1 | 2 | 3 | 9
    Probable UIP pattern HRCT scan prior to screening. Lung biopsy in accordance with HRCT: NA | 3 | 1 | 2 | 3 | 9
    Probable UIP pattern HRCT scan prior to screening. Lung biopsy in accordance with HRCT: YES: number analyzed (Participants) | 3 | 1 | 2 | 3 | 9
    Probable UIP pattern HRCT scan prior to screening. Lung biopsy in accordance with HRCT: YES | 0 | 1 | 1 | 2 | 4
Antifibrotic treatment for IPF [Count of Participants; unit: Participants]
  NO | 2 | 4 | 4 | 2 | 12
  YES | 4 | 2 | 2 | 4 | 12
  Nintedanib | 3 | 2 | 1 | 3 | 9
  Pirfenidone | 1 | 0 | 1 | 1 | 3
Number of subjects with no exacerbations in the 3 months before screening [Count of Participants; unit: Participants] — The measure shows the number of subjects with 0 exacerbations.
  Participants | 6 | 6 | 6 | 6 | 24
FEV1 actual value [Mean (Standard Deviation); unit: liters] | 2.190 (0.343) | 2.550 (0.735) | 2.107 (0.628) | 2.405 (0.308) | 2.313 (0.530)
FEV1 % of predicted [Mean (Standard Deviation); unit: % of predicted normal value] | 69.90 (11.28) | 85.75 (15.97) | 77.67 (13.64) | 81.05 (10.74) | 78.59 (13.55)
FVC actual value [Mean (Standard Deviation); unit: liters] | 2.818 (0.385) | 3.267 (1.116) | 2.632 (0.914) | 2.965 (0.429) | 2.920 (0.762)
FVC % of predicted normal value [Mean (Standard Deviation); unit: % of predicted normal value] | 70.33 (13.17) | 85.23 (20.15) | 75.67 (14.11) | 75.72 (10.57) | 76.74 (14.95)

OUTCOME MEASURES:

1. Primary Outcome: 1_Subjects With Adverse Event (AE); Non-Serious AEs and Serious AEs
Description: Evaluate reported adverse events (AEs) and serious adverse events (SAEs). The number of subjects affected by AEs or SAEs is presented below.
  Please note: comprehensive summaries of AEs and SAEs are presented in section 'Adverse Events'; these include the preferred term of the AE or SAE, the number of subjects affected, and the number of events for a each preferred term.
Time Frame: From pre-dose (baseline) up to day 84.
Population: Safety set: all randomised subjects who received a dose of study treatment, including partial dose.
Measure: Count of Participants; unit: Participants
Arm/Group | CHF 10067 1000 mg (Test Treatment) | CHF 10067 2000 mg (Test Treatment) | CHF 10067 3000 mg (Test Treatment) | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6
Participants
  Serious TEAE | 0 | 0 | 1 | 0
  Non-serious TEAE | 4 | 3 | 5 | 4
  AE leading to study treatment discontinuation | 0 | 0 | 0 | 0
  AE leading to death | 0 | 0 | 0 | 0

2. Secondary Outcome: 2_Systemic Exposure [Area Under the Concentration-time Curve From Zero to Time (AUC0-t)]
Description: Evaluate the area under the concentration-time curve (AUC) from zero to the last quantifiable concentration (AUC0-t) of CHF10067 after a single dose.
Time Frame: Pre-dose (within 75 min from start of infusion, baseline), at the end of infusion, 2, 4, 8, and 20 h after the end of infusion and 5, 7, 14, 28, 56, and 84 days post-dose.
Population: Pharmacokinetic set (PK set): all subjects from the safety set, excluding subjects without any valid PK measurement or with important protocol deviations significantly affecting PK, for example, use of non-permitted medications.
Measure: Mean (Standard Deviation); unit: day.μg/mL
Arm/Group | CHF 10067 1000 mg (Test Treatment) | CHF 10067 2000 mg (Test Treatment) | CHF 10067 3000 mg (Test Treatment)
Number analyzed (Participants) | 6 | 6 | 6
day.μg/mL | 3424 (647) | 7902 (1001) | 15592 (3027)

3. Secondary Outcome: 3_Area Under the Concentration-time Curve (AUC) From Zero to Infinity (AUC0-∞)
Description: Evaluate the area under the concentration-time curve (AUC) from zero to infinity (AUC0-∞) of CHF10067 after a single dose.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: day.μg/mL
Arm/Group | CHF 10067 1000 mg (Test Treatment) | CHF 10067 2000 mg (Test Treatment) | CHF 10067 3000 mg (Test Treatment)
Number analyzed (Participants) | 6 | 6 | 6
day.μg/mL | 3450 (660) | 8141 (1112) | 16328 (3245)

4. Secondary Outcome: 4_Pharmacokinetics -- Maximum Plasma Concentration (Cmax)
Description: Evaluate the Cmax (maximum observed concentration) after a single dose of CHF10067.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | CHF 10067 1000 mg (Test Treatment) | CHF 10067 2000 mg (Test Treatment) | CHF 10067 3000 mg (Test Treatment)
Number analyzed (Participants) | 6 | 6 | 6
μg/mL | 307 (43.9) | 668 (126) | 1067 (173)

5. Secondary Outcome: 5_Pharmacokinetics -- Time to Maximum Observed Concentration (Tmax)
Description: Evaluate the time to maximum observed concentration (tmax).
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Median (Full Range); unit: hour
Arm/Group | CHF 10067 1000 mg (Test Treatment) | CHF 10067 2000 mg (Test Treatment) | CHF 10067 3000 mg (Test Treatment)
Number analyzed (Participants) | 6 | 6 | 6
hour | 1.69 [1.67 to 3.67] | 3.78 [3.58 to 11.67] | 5.39 [5.35 to 7.43]

6. Secondary Outcome: 6_Pharmacokinetics -- Serum Concentration at the End of Infusion (Cinf)
Description: Evaluate serum concentration at the end of infusion (Cinf) of CHF10067.
Time Frame: Pre-dose (within 75 min from start of infusion, baseline), at the end of infusion (up to 6 hours from the start of infusion).
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | CHF 10067 1000 mg (Test Treatment) | CHF 10067 2000 mg (Test Treatment) | CHF 10067 3000 mg (Test Treatment)
Number analyzed (Participants) | 6 | 6 | 6
μg/mL | 304 (44.6) | 658 (138) | 1065 (174)

7. Secondary Outcome: 7_Pharmacokinetics -- Time at the End of Infusion (Tinf)
Description: Evaluate the time of serum concentration at the end of infusion (Tinf). Time at the end of the infusion.
Time Frame: as for outcome 6
Population: as for outcome 2
Measure: Median (Full Range); unit: hour
Arm/Group | CHF 10067 1000 mg (Test Treatment) | CHF 10067 2000 mg (Test Treatment) | CHF 10067 3000 mg (Test Treatment)
Number analyzed (Participants) | 6 | 6 | 6
hour | 1.68 [1.67 to 1.72] | 3.69 [3.58 to 3.85] | 5.38 [5.35 to 5.50]

8. Secondary Outcome: 8_Pharmacokinetics -- Clearance (CL)
Description: Evaluate clearance (CL) of CHF10067.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: liter/day
Arm/Group | CHF 10067 1000 mg (Test Treatment) | CHF 10067 2000 mg (Test Treatment) | CHF 10067 3000 mg (Test Treatment)
Number analyzed (Participants) | 6 | 6 | 6
liter/day | 0.295 (0.0489) | 0.250 (0.0357) | 0.190 (0.0363)

9. Secondary Outcome: 9_Pharmacokinetics -- Volume of Distribution (Vz)
Description: Evaluate volume of distribution (Vz) CHF10067.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: liter
Arm/Group | CHF 10067 1000 mg (Test Treatment) | CHF 10067 2000 mg (Test Treatment) | CHF 10067 3000 mg (Test Treatment)
Number analyzed (Participants) | 6 | 6 | 6
liter | 4.93 (0.969) | 5.99 (0.716) | 5.21 (1.03)

10. Secondary Outcome: 10_Pharmacokinetics -- Terminal Half-life (t1/2)
Description: Evaluate the terminal half-life (t1/2) of CHF10067.
Time Frame: From pre-dose (baseline) up to day 84.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: days
Arm/Group | CHF 10067 1000 mg (Test Treatment) | CHF 10067 2000 mg (Test Treatment) | CHF 10067 3000 mg (Test Treatment)
Number analyzed (Participants) | 6 | 6 | 6
days | 11.7 (2.20) | 16.8 (2.32) | 19.1 (1.93)

11. Secondary Outcome: 11_Spirometry -- Forced Expiratory Volume in the First Second (FEV1) -- Percent Predicted -- Change From Baseline
Description: Forced expiratory volume in the first second (FEV1) parameters, summarised using descriptive statistics at each analysis time point by treatment.
  Summary results show the change from baseline of the percent predicted.
Time Frame: Pre-dose (baseline), and on 7, 28, 56, and 84 day post-dose.
Population: Safety set: all subjects who were randomised and received a dose of study treatment, including partial dose.
Measure: Mean (Standard Deviation); unit: percent predicted FEV1
Arm/Group | CHF 10067 1000 mg (Test Treatment) | CHF 10067 2000 mg (Test Treatment) | CHF 10067 3000 mg (Test Treatment) | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6
percent predicted FEV1
  Day 7 | 3.93 (3.35) | 0.50 (2.74) | -0.20 (1.34) | -0.43 (2.60)
  Day 28: number analyzed (Participants) | 5 | 6 | 6 | 6
  Day 28 | 3.76 (3.66) | -0.55 (3.06) | -2.93 (2.81) | -0.55 (3.37)
  Day 56: number analyzed (Participants) | 5 | 6 | 6 | 6
  Day 56 | 3.18 (3.58) | -0.68 (3.54) | -0.75 (5.68) | -1.35 (2.93)
  Day 84: number analyzed (Participants) | 6 | 5 | 6 | 6
  Day 84 | 0.13 (5.57) | 0.36 (4.30) | -2.70 (2.93) | -1.40 (3.62)

12. Secondary Outcome: 12_Spirometry -- Forced Vital Capacity (FVC) -- Percent Predicted -- Change From Baseline
Description: Forced vital capacity (FVC) parameters will be summarised using descriptive statistics at each analysis time point by treatment.
  Summary results show the change from baseline of the percent predicted.
Time Frame: Text adjusted Pre-dose (baseline), and on 7, 28, 56, and 84 day post-dose.
Population: Safety set: all subjects who were randomised and received a dose of study treatment, including partial dose.
Measure: Mean (Standard Deviation); unit: percent predicted FVC
Arm/Group | CHF 10067 1000 mg (Test Treatment) | CHF 10067 2000 mg (Test Treatment) | CHF 10067 3000 mg (Test Treatment) | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6
percent predicted FVC
  Day 7 | 3.12 (2.24) | -0.90 (3.31) | -0.50 (2.89) | -0.92 (3.80)
  Day 28: number analyzed (Participants) | 5 | 6 | 6 | 6
  Day 28 | 2.70 (3.74) | -0.50 (2.58) | -3.23 (2.76) | -0.13 (4.10)
  Day 56: number analyzed (Participants) | 5 | 6 | 5 | 6
  Day 56 | 2.50 (1.87) | -1.17 (3.12) | -1.42 (6.55) | -0.90 (2.84)
  Day 84: number analyzed (Participants) | 6 | 5 | 6 | 6
  Day 84 | -0.72 (4.02) | -0.36 (3.56) | -1.98 (3.79) | -1.97 (3.22)

13. Secondary Outcome: 13_Vital Signs -- Abnormal Changes in Systolic and Diastolic Blood Pressure
Description: Evaluate abnormal changes in systolic and diastolic blood pressure from baseline at any post-baseline time point.
Time Frame: From pre-dose (baseline) up to day 84.
Population: Safety set: all subjects who were randomised and received a dose of study treatment, including partial dose.
Measure: Count of Participants; unit: Participants
Arm/Group | CHF 10067 1000 mg (Test Treatment) | CHF 10067 2000 mg (Test Treatment) | CHF 10067 3000 mg (Test Treatment) | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6
Participants
  Systolic Blood Pressure Decrease From Baseline >20 mmHg | 3 | 0 | 1 | 2
  Systolic Blood Pressure Increase From Baseline >20 mmHg | 1 | 0 | 1 | 2
  Diastolic Blood Pressure Decrease From Baseline >10 mmHg | 3 | 5 | 5 | 4
  Diastolic Blood Pressure Increase From Baseline >10 mmHg | 2 | 2 | 2 | 3

14. Secondary Outcome: 14_Immunogenicity Profile -- Anti-drug Antibody (ADA) and Neutralising Antibody (nAb).
Description: Evaluate the immunogenicity profile of CHF 10067 in serum, with respect to the development of anti-drug antibody (ADA) and neutralising antibody (nAb).
  A robust immunogenicity profile indicates the potential for the drug to trigger an immune response in patients, leading to the formation of ADAs. These antibodies can affect the drug's efficacy, safety, and pharmacokinetics.
  Detecting the presence of ADAs in serum samples was performed using an enzyme linked immunosorbent assay (ELISA), a validated assay method. Neutralizing Antibody (nAb) are a subset of ADAs that can interfere with the drug's therapeutic activity by blocking its binding to the target or inhibiting its downstream effects. The presence of ADAs and nAbs can affect the drug's pharmacokinetics (PK) by altering its absorption, distribution, metabolism, and excretion. This can lead to changes in drug exposure and potentially impact efficacy and safety.
Time Frame: Pre-dose (baseline), at day 14, 28, 56, 84, and in case of early termination.
Population: Safety set: all subjects who were randomised and received a dose of study treatment, including partial dose.
Measure: Count of Participants; unit: Participants
Arm/Group | CHF 10067 1000 mg (Test Treatment) | CHF 10067 2000 mg (Test Treatment) | CHF 10067 3000 mg (Test Treatment) | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6
Participants
  1_Baseline ADA positive | 0 | 0 | 0 | 0
  2_ADA prevalence | 1 | 0 | 0 | 0
  3_ADA incidence (ADA+) | 1 | 0 | 0 | 0
  4_Duration of ADA Persistently positive ADA | 0 | 0 | 0 | 0
  5_Duration of ADA Transiently positive ADA | 1 | 0 | 0 | 0
  6_Treatment-boosted ADA | 0 | 0 | 0 | 0
  7_nAb positive at any visit | 1 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events (AE) were reported from the time of patient informed consent signature until subject's study participation ended (day 84 or early withdrawal).
Description: Analyses of safety parameters were based on the safety set, defined as all subjects who were randomised and received a dose of study treatment, including partial dose.
  Adverse events were analysed according to the treatment-emergent principle.
  The end of the study was defined as the last visit of the last subject in the study.
Arm/Group | CHF 10067 1000 mg (Test Treatment) | CHF 10067 2000 mg (Test Treatment) | CHF 10067 3000 mg (Test Treatment) | Placebo
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 1/6 | 0/6
Other Adverse Events (participants affected / at risk) | 4/6 | 3/6 | 5/6 | 4/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CHF 10067 1000 mg (Test Treatment) (N=6) | CHF 10067 2000 mg (Test Treatment) (N=6) | CHF 10067 3000 mg (Test Treatment) (N=6) | Placebo (N=6)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CHF 10067 1000 mg (Test Treatment) (N=6) | CHF 10067 2000 mg (Test Treatment) (N=6) | CHF 10067 3000 mg (Test Treatment) (N=6) | Placebo (N=6)
Supraventricular Extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Periorbital Oedema (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (4)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Fatigue (General disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Medical Device Site Rash (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lower Respiratory Tract Infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Tinea Pedis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin Abrasion (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Blood Creatinine Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (3)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Sputum Discoloured (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dry Skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Results of this study may be published or presented at scientific meetings. If a publication is presented by the Investigator, the Investigator agrees to submit all manuscripts or abstracts to the Sponsor to Chiesi before submission.

DOCUMENTS (2):
  • Study Protocol (2023-07-06): https://cdn.clinicaltrials.gov/large-docs/50/NCT05513950/Prot_000.pdf
  • Statistical Analysis Plan (2024-05-30): https://cdn.clinicaltrials.gov/large-docs/50/NCT05513950/SAP_001.pdf